CLINICAL TRIAL: NCT01864551
Title: Comparison of Olanzapine and Lamotrigine in the Prevention of Recurrence of Depressive Episode in the Patients With Bipolar Disorders
Brief Title: Olanzapine Compared to Lamotrigine in the Prevention of Depressive Episode in the Patients With Bipolar Disorder
Acronym: OCTLPODEPWBD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Chin-Bin Yeh, Attending Physician, Tri-Service General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TSGH 097-05-061
Record Dates: First submitted 2013-05-03; First posted 2013-05-29 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Lamotrigine; Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- lamotrigine (Active Comparator): maintenance treatment of the patients with bipolar disorder with olanzapine or lamotrigine
  Interventions: Drug: Lamotrigine
- olanzapine (Active Comparator): maintenance treatment of the patients with bipolar disorder with olanzapine or lamotrigine
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Lamotrigine
  Other Names: lamictal
  Arms: lamotrigine
Drug: Olanzapine
  Arms: olanzapine

SUMMARY:
The investigators hypothesized that olanzapine will be superior to lamotrigine in the prevention of any kind of recurrence of bipolar disorder. On the other hand, lamotrigine group will have better prevention of depressive episode than olanzapine group. Meanwhile, the investigators supposed that there will be more concomitant medicine in lamictal group than olanzapine group. The comorbidity will influence the measurement of outcome such as time period of recurrence of depressive episode in both groups..

DETAILED DESCRIPTION:
Background:

Bipolar disorder is a highly recurrent disease and has great impact on the function of patients. Depressive symptoms consist of more than 50% of life time during the illness and may lead to self harm or suicidal behaviors. Lamotrigine, a kind of mood stabilizer, was proved to be effective in preventing depressive episode in Bipolar disorder. However, it is still lacking evidence that monotherapy with atypical antipsychotics such as olanzapine had the efficacy of preventing the recurrence of depressive episode in the patients with bipolar disorder although it had demonstrated good prevention in manic episode of bipolar disorder.

Methods:

The investigators will enroll 60 patients who had bipolar disorder in remission state for at least two months and have already received olanzapine or lamotrigine as the maintenance treatment. The patients maintained with olanzapine will be applied to olanzapine group (N=30) whereas those maintained on lamotrigine will be applied to lamotrigine group (N=30) for one month before entering into this study. They will be followed up to 12 months. The demography data will be compared between two groups. The concomitant medicine in the maintenance period of the subjects recruited will be recorded and analyzed. The time period to recurrence of depressive episode will be compared between groups. In addition, they will investigate if there is any independent factor such as comorbid substance use disorder, alcohol use disorder, personality disorders, other psychiatric disorders (posttraumatic stress disorder, eating disorder), or medical illness correlating with higher recurrent rate of depressive episode in bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

The patients aged 15 to 50 who have bipolar disorder defined by the DSM-IV in remission state(YMRS<12, HAMD<7, CDR<3) for at least two months and have already received olanzapine or lamotrigine as the maintenance treatment for one month. In addition, they should have at least three hypomanic, manic, depressive or mixed episodes previously.

Exclusion Criteria:

1. The patients are not willing to participate in the study after detailed explanation.
2. The patients who could not followed the investigators' instruction
3. The patients who have severe neurological or mental illness like epileptic disorder, history of stroke, schizophrenia, schizoaffective disorder, mental retardation or uncontrolled suicide risk.
4. The patients who have severe medical illness or surgical conditions like uncontrolled abnormal thyroid function, history of heart attack, uncontrolled hypertension.
5. The patient who are taking other mood stabilizers or antipsychotics within one month prior to the evaluation of entering our study.
6. The patients who are taking medications that might interfere with the metabolism of olanzapine or lamotrigine.
7. The patient who are allergy to olanzapine or lamotrigine.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2008-08; Primary Completion 2009-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
time period to the recurrence of depressive episode | 12 months
  comparison of the time period to recurrent depressive episode between two groups

SECONDARY OUTCOMES:
the recurrent depressive episode | 12 months
  if there is any depressive episode during follow-up period

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Pan PY, Lee MS, Lo MC, Yang EL, Yeh CB. Olanzapine is superior to lamotrigine in the prevention of bipolar depression: a naturalistic observational study. BMC Psychiatry. 2014 May 19;14:145. doi: 10.1186/1471-244X-14-145. PMID 24885966